CLINICAL TRIAL: NCT00696579
Title: BCG vs. Gemcitabine For Intravesical Therapy In High Risk Superficial Bladder Cancer: A Randomized Prospective Study
Brief Title: Bacillus of Calmette and Guerin (BCG) Versus Gemcitabine For Intravesical Therapy In High Risk Superficial Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Of Perugia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC_ML_003
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Bladder Cancer
Keywords: BCG; Gemcitabine; Intravesical; Therapy; Superficial; Transitional; Cell carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Group A received BCG instillation 14 days after II look-TURB:6 weekly instillations of Tice-strain BCG (Organon Teknika Corp.) as induction chemotherapy, with a dose of 5 x 108 CFU diluted in 50 mL of saline held in the bladder for 2 hours.
  Interventions: Drug: BCG
- 2 (Experimental): 14 days after II look-TURB the patients received 6 weekly instillations of Gemcitabine (Gemzar, Eli Lilly SpA), using a dose of 2000 mg diluted in 50 mL of saline held in the bladder for 2 hours
  Interventions: Drug: gemcitabine

INTERVENTIONS:
Drug: BCG — 6 weekly instillations of Tice-strain BCG (Organon Teknika Corp.) as induction chemotherapy, with a dose of 5 x 108 CFU diluted in 50 mL of saline held in the bladder for 2 hours.
  Arms: A
Drug: gemcitabine — 14 days after II look-TURB the patients received 6 weekly instillations of Gemcitabine (Gemzar, Eli Lilly SpA), using a dose of 2000 mg diluted in 50 mL of saline held in the bladder for 2 hours
  Arms: 2

SUMMARY:
A significant number of patients with high risk superficial bladder cancer has progression to invasive disease. No consensus exists regarding the optimal treatment to decrease the recurrence and progression rate. The aim of this research is to evaluate the safety, tolerability and efficacy of adjuvant intravesical gemcitabine vs. BCG in the treatment of high-risk superficial bladder cancer

DETAILED DESCRIPTION:
This was a prospective, randomized study conducted from 2004 to 2006 at a single tertiary urban teaching University Urological Department regarding sixty-four patients with high-risk superficial bladder cancer (pT1, and/or G3 and/or CIS), who were assigned to interventions (gemcitabine or BCG) by using random allocation 1:1. Group A, 32 patients, were treated weekly (6 weekly instillations) with BCG dose 5 x 108 CFU and then maintenance therapy at 3-6-12-18-24-30-36 months; Group B, 32 patients, received gemcitabine 2 gr/instillation on a weekly basis (6 weekly instillations), followed by maintenance therapy at 3-6-12-18-24-30-36 months.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of high risk superficial bladder cancer according to EAU guidelines (http://www.eortc.be/tools/bladdercalculator/),
* Having never been treated with other intravesical chemotherapeutic agents,
* And to consent to participate to the study

Exclusion Criteria:

* Concomitant tumours;
* Urinary tract infections (UTI);
* Altered function of the liver, kidneys and/or bone marrow;
* Major cardiovascular diseases;
* Life expectancy of less than 1 year;
* Intravesical chemotherapy in the previous 3 months or immunotherapy in the previous 6 months;
* Systemic chemotherapy and pelvic radiotherapy prior to TURB, and any condition that in the judgment of the investigators would interfere with the subject's ability to provide informed consent, comply with study instructions, place the subject at increased risk, or which might confound interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-01; Primary Completion 2008-03

PRIMARY OUTCOMES:
The primary outcome measure consists of evaluation of recurrence and progression rates as they were detected by follow-up tools. Interval before recurrence and progression were also considered primary end-points

SECONDARY OUTCOMES:
Secondary endpoints were tolerability, as detected by number of patients who dropped out the study, and safety as the recording of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- 1. Department of Medical-Surgical Specialties and Public Health, Section of Urology and Andrology, University of Perugia - Italy, Perugia, Italy